CLINICAL TRIAL: NCT02640443
Title: Sulfamethoxazole for the Treatment of Primary PREPL Deficiency (In Dutch: Sulfamethoxazole Ter Behandeling Van Primaire PREPL deficiëntie)
Brief Title: Sulfamethoxazole for the Treatment of Primary PREPL Deficiency
Acronym: SPPD
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Universitair Ziekenhuis Brussel (Other)
Collaborators: KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 2015/059
Record Dates: First submitted 2015-10-07; First posted 2015-12-29 (Estimated); Last update posted 2015-12-29 (Estimated); Status verified 2015-10

CONDITIONS: Hypotonia Cystinuria Syndrome; Isolated PREPL Deficiency
MeSH Terms: conditions — Hypotonia-Cystinuria Syndrome | interventions — Sulfamethoxazole

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): Treatment with sulfamethoxazole. Subjects will serve as their own control, by using the data from baseline and after treatment stop.
  Interventions: Drug: Sulfamethoxazole

INTERVENTIONS:
Drug: Sulfamethoxazole — 60 mg sulfamethoxazole per kg bodyweight (maximal of 3g) divided in 2 doses per day during 3 weeks

SUMMARY:
The investigators will evaluate whether sulfamethoxazole, a sulfamide antibiotic, improves the symptoms of primary PREPL deficiency (hypotonia-cystinuria syndrome and isolated PREPL deficiency).

ELIGIBILITY:
Inclusion Criteria:

* patients with molecular confirmation of primary PREPL deficiency
* who are able to follow the study protocol (for the primary endpoint)
* who have given written informed consent

Exclusion Criteria:

* age<2m
* women of child-bearing age unless using a reliable method for contraception and not pregnant at study entrance
* additional diagnosis with influence on muscle force
* not able to follow the study protocol (for the primary endpoint)
* history of sulfonamide hypersensitivity
* diminished renal function based on serum creatinine
* transaminases higher than 3 times the upper limit of normal
* for the pupillometry: eye pathology with the exception of refractive errors, drugs with influence on the pupillary light reflex

Min Age: 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-10 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Change in ptosis on myasthenia gravis composite scale | Change in score between baseline/1 week after treatment stop versus third week of treatment
  ptosis item on the myasthenia gravis composite scale: single blinded scoring on video-images
Change in ptosis index | Change in index between baseline/1 week after treatment stop versus third week of treatment
  ptosis index, single blinded measurement on photograph
Change in lip length index | Change in index between baseline/1 week after treatment stop versus third week of treatment
  lip length index, single blinded measurement on photographs
Change in lip purse index | Change in index between baseline/1 week after treatment stop versus third week of treatment
  Lip purse index, single blinded measurement on photographs

SECONDARY OUTCOMES:
Change in satiety | Change in Composite score between baseline/1 week after treatment stop versus third week of treatment
  satiety scale (visual analog); 4 questions are asked, a compositie score is made, by adding the different scores (the answers on questions 2 and 3 are counted as negative values)
Change in myasthenia gravis composite score | Change in score between baseline/1 week after treatment stop versus third week of treatment
  Sum of all the subscores
myasthenia gravis composite dysarthria and eye closure subscores | Change in score between baseline/1 week after treatment stop versus third week of treatment
  scored on video
Change in muscle strength | Change in strength between baseline/1 week after treatment stop versus third week of treatment
  scored with hand-held manometry
Change in complete blood count | Change between baseline/1 week after treatment stop versus third week of treatment
  complete blood count (development of cytopenia)
Change in Glycemia | Change between baseline/1 week after treatment stop versus third week of treatment
  Glycemia
Change in renal ultrasound | development of kidney stones after the third week of treatment versus baseline
  renal ultrasound
Change in myasthenia gravis-activities of daily life | Change in score between baseline/1 week after treatment stop versus third week of treatment
  Scale with rating of activities of daily life
Change in neuropsychology Child Behaviour checklist | Change in score between baseline/1 week after treatment stop versus third week of treatment
  composite score of Child Behaviour checklist
Change in neuropsychology Brief | Change in score between baseline/1 week after treatment stop versus third week of treatment
  composite score of Brief
Change in neuropsychology Amsterdamse neuropsychologische test | Change in score between baseline/1 week after treatment stop versus third week of treatment
  composite score of Amsterdamse Neuropsychologische test (ANT)
Change in Insulin | Change between baseline/1 week after treatment stop versus third week of treatment
  insulin
Change in IGF1 | Change between baseline/1 week after treatment stop versus third week of treatment
  IGF-1
Change in IGFPB3 | Change between baseline/1 week after treatment stop versus third week of treatment
  IGFBP3
Change in pupillometry | Change between baseline/1 week after treatment stop versus third week of treatment
  dynamic pupillometry with infrared camera

CONTACTS AND LOCATIONS:
Overall Officials: Luc Régal, MD, Principal Investigator — Universitair Ziekenhuis Brussel

REFERENCES:
- [Background] Regal L, Shen XM, Selcen D, Verhille C, Meulemans S, Creemers JW, Engel AG. PREPL deficiency with or without cystinuria causes a novel myasthenic syndrome. Neurology. 2014 Apr 8;82(14):1254-60. doi: 10.1212/WNL.0000000000000295. Epub 2014 Mar 7. PMID 24610330